CLINICAL TRIAL: NCT01165476
Title: An Evaluation of the Comparative Bioavailability of a Single Oral Dose of 1mg UT-15C (Treprostinil Diethanolamine) SR Tablets Manufactured by Two Independent Facilities Administered to Healthy Volunteers in the Fed State
Brief Title: Comparative Bioavailability of Treprostinil Diethanolamine Manufactured by Two Independent Facilities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Andrew Nelsen, PharmD, United Therapeutics
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-121
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: treprostinil; bioavailability; bioequivalence
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- manufacturer #1 (Active Comparator): treprostinil diethanolamine from manufacturer #1
  Interventions: Drug: Treprostinil diethanolamine
- manufacturer #2 (Experimental): treprostinil diethanolamine from manufacturer #2
  Interventions: Drug: Treprostinil diethanolamine

INTERVENTIONS:
Drug: Treprostinil diethanolamine — sustained release tablets. One 1mg tablet per period. Two total doses.

SUMMARY:
The purpose of this study is to compare the bioavailability of a single 1mg dose of treprostinil diethanolamine sustained release (SR) tablets manufactured by two independent facilities.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy and between the ages of 18 and 55 years, inclusive, at Screening
* Female subjects must weigh between 45 and 100 kg, inclusive, with a BMI between 19.0-29.9 kg/m2, inclusive at Screening. Male subjects must weigh between 50 and 120 kg, inclusive, with a BMI between 19.0-32.0 kg/m2, inclusive at Screening
* Subject has a medical history, physical examination, vital signs, ECG and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at Screening

Exclusion Criteria:

* Subject has any clinically relevant abnormality identified during the screening physical examination, 12-lead ECG, or laboratory examinations.
* Subject has a history of anaphylaxis, a documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug
* Subject has a clinically significant history of neurological, cardiovascular,respiratory, endocrine, hematological, hepatic, renal, gastrointestinal,genitourinary, pulmonary, and/or musculoskeletal disease; glaucoma; a psychiatric disorder, or any other chronic disease, whether controlled by medication or not.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Treprostinil pharmacokinetics | 36 hours
  Treprostinil pharmacokinetics in healthy volunteers following a single oral dose of 1mg treprostinil diethanolamine collecting pre and post-dose levels to 36 hours.

SECONDARY OUTCOMES:
Clinical lab values | Days 0, 7 and 9
Adverse event monitoring | From signing of ICF to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Aziz L Laurent, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, Austin, Texas, United States